CLINICAL TRIAL: NCT04287426
Title: A Single-blinded Multicenter Randomized Study Comparing Intubating Conditions After Either Rocuronium 0.6 mg/kg or Remifentanil 2 µg/kg in Elderly Patients
Brief Title: A Comparison of Rocuronium 0.6 mg/kg and Remifentanil 2 µg/kg in Elderly Patients Over 80 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Matias Vested, Principal Investigator, Anesthesiologist, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-19070343; 2019-004121-25 (EudraCT Number)
Record Dates: First submitted 2020-01-27; First posted 2020-02-27 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Neuromuscular Blockade; Intubation Complication; Anesthesia
MeSH Terms: interventions — Rocuronium; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receiving rocuronium at induction (Active Comparator): Rocuronium 0,6 mg/kg at induction
  Interventions: Drug: Rocuronium 0.6 mg/kg
- Group receiving remifentanil at induction (Active Comparator): Remifentanil 2 μg/kg at induction
  Interventions: Drug: Remifentanil 2 µg/kg

INTERVENTIONS:
Drug: Rocuronium 0.6 mg/kg — Rocuronium 0.6 mg/kg is compared to patients with 2 µg/kg remifentanil
  Arms: Group receiving rocuronium at induction
Drug: Remifentanil 2 µg/kg — Rocuronium 0.6 mg/kg is compared to patients with 2 µg/kg remifentanil
  Arms: Group receiving remifentanil at induction

SUMMARY:
The number of elderly patients above 80 years is increasing and a large proportion of these patients will require surgery and anesthesia.

During anesthesia neuromuscular blocking agents (NMBA) are administered to facilitate intubating conditions and reduce the trauma to the larynx and vocal cords. There is a risk of residual neuromuscular block when using NMBAs like rocuronium.

Remifentanil is a fentanyl analogue commonly used for induction since it also facilitates intubation. There is no risk of residual neuromuscular block, nonetheless circulatory side effects have been seen.

It is unknown which is superior concerning intubating conditions in elderly patients. Therefore, the aim of this study is to determine the effect on intubating conditions and laryngeal morbidity after either rocuronium 0.6 mg/kg or remifentanil 2 µg/kg in patients with age ≥ 80 years. The hypothesis of this study is that rocuronium 0.6 mg/kg provides a higher proportion with excellent intubating conditions compared to remifentanil 2 µg/kg.

DETAILED DESCRIPTION:
The number of elderly patients (>80 years) is increasing and a large proportion of these patients will require surgery and anesthesia within the next decades. Elderly patients are at higher risk of major morbidity and mortality and are characterized by a reduction in cardiac output, liver function and renal function. These physiological changes influence pharmacodynamics and pharmacokinetics of drugs administered during anesthesia.

During anesthesia neuromuscular blocking agents (NMBA) are administered to facilitate intubating conditions and reduce the trauma to the larynx and vocal cords. Studies suggests that avoidance of neuromuscular blocking agents (NMBAs) increases the risk of difficult tracheal intubation and leads to impaired intubating conditions with direct laryngoscopy. Furthermore, avoidance of NMBA significantly increases the risk of upper airway discomfort or injury. Even low doses of rocuronium may be associated with a significant improvement of intubating conditions.

Remifentanil is a fentanyl analogue commonly used for induction since it also facilitates intubation. There is no risk of residual neuromuscular block, nonetheless circulatory side effects have been seen.

The possible benefit in this trial is to investigate whether rocuronium 0.6 mg/kg or remifentanil 2 µg/kg provides best intubating conditions in the elderly. This may result in different intubating difficulty scores between the two groups of elderly patients. The results may help to detect the optimal method for intubation of the trachea in elderly patients.

The aim of this study is to determine the effect on intubating conditions and laryngeal morbidity after either rocuronium 0.6 mg/kg or remifentanil 2 µg/kg in patients with age ≥ 80 years. The hypothesis of this study is that rocuronium 0.6 mg/kg provides a higher proportion with excellent intubating conditions compared to remifentanil 2 µg/kg.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 80
* Scheduled for elective operations (expected duration of anesthesia > 1 hour) under general anesthesia with intubation
* American Society of Anesthesiologists physical status classification (ASA) I to III
* Informed consent (see appendix 1)
* Read and understand Danish

Exclusion Criteria:

* Neuromuscular disease
* Known allergy to rocuronium, remifentanil or sugammadex
* Rapid sequence induction

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-13 (Actual)

PRIMARY OUTCOMES:
Evaluation of intubating conditions ad modum Fuchs-Buder et al | 2 minutes after start of administration of trial medication
  Occurrence of excellent intubating conditions 2 minutes after start of administration of 0.6 mg/kg rocuronium or 2 µg/kg remifentanil, scored according to Fuchs-Buder et al. The intubating conditions will be classified as excellent if all qualities are excellent, good if all qualities are either excellent or good and poor if the presence of a single quality is listed as poor.

SECONDARY OUTCOMES:
Subjective side effects of laryngoscopy | 24 hours postoperatively and 3 days postoperatively
  After 24 hours patients are asked about hoarseness and sore throat. The patients who experience either or both will be called 3 days postoperatively again. These two variables are assessed using a numeric ranking scale.
Dose of ephedrine or dose of metaoxedrine administered | From induction until the patient is ready to be positioned for surgery, ranging from 5 minutes up to 1 hour.
  If ephedrine and/or metaoxedrine is administered in the time period from induction until the patient is ready to be positioned for surgery it will be noted in the CRF. The amount administered will also be noted in the CRF. Changes in blood pressure are treated according to local guidelines.
Intubating conditions according to IDS | 2 minutes after start of administration of trial medication
  Another way of rating intubating conditions are by an intubating difficulty scale (Table 2) (20) 2 minutes after injection of rocuronium/remifentanil. The investigator performing the intubation will be handed the CRF where he/she will fill out Table 2. Furthermore, investigator will note if a stylet or video laryngoscope has been used.

CONTACTS AND LOCATIONS:
Overall Officials: Matias Vested, MD, PhD, Principal Investigator — Department of Anaesthesia, Head and Orthopaedics Centre, Rigshospitalet, Denmark; Anne Marie Sørensen, MD, PhD, Principal Investigator — Department of Neuroanaesthesia, Rigshospitalet, Glostrup, Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Rigshospitalet, Glostrup, Glostrup Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vested M, Sorensen AM, Bjerring C, Christensen RE, Dinesen F, Vang M, Gilvanoff A, Hansen TE, Nielsen T, Rasmussen LS. A blinded randomized study comparing intubating conditions after either rocuronium 0.6 mg.kg-1 or remifentanil 2 microg.kg-1 in elderly patients. Acta Anaesthesiol Scand. 2021 Nov;65(10):1367-1373. doi: 10.1111/aas.13957. Epub 2021 Sep 5. PMID 34310692